CLINICAL TRIAL: NCT07283263
Title: A Phase 1, Randomized, Placebo-Controlled, Double-Blind, First-in-Human Study Evaluating Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of Orally Administered BMS-986521 in Healthy Adult Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, and Drug Levels of BMS-986521 in Healthy Participants.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CN014-0001
Record Dates: First submitted 2025-12-02; First posted 2025-12-15 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Pharmacokinetics; BMS-986521; Placebo; Drug-food Interaction; Single Ascending Dose (SAD); Multiple Ascending Dose (MAD); Elderly; Relative Bioavailability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Part A Cohort 1 (Experimental)
  Interventions: Drug: BMS-985521; Other: Placebo
- Part A Cohort 2 (Experimental)
  Interventions: Drug: BMS-985521; Other: Placebo
- Part A Cohort 3 (Experimental)
  Interventions: Drug: BMS-985521; Other: Placebo
- Part A Cohort 4 (Experimental)
  Interventions: Drug: BMS-985521; Other: Placebo
- Part A Cohort 5 (Experimental)
  Interventions: Drug: BMS-985521; Other: Placebo
- Part A Cohort 6 (Experimental)
  Interventions: Drug: BMS-985521; Other: Placebo
- Part B Cohort 7 (Experimental)
  Interventions: Drug: BMS-985521; Other: Placebo
- Part B Cohort 8 (Experimental)
  Interventions: Drug: BMS-985521; Other: Placebo
- Part B Cohort 9 (Experimental)
  Interventions: Drug: BMS-985521; Other: Placebo
- Part B Cohort 10 (Experimental)
  Interventions: Drug: BMS-985521; Other: Placebo
- Part B Cohort 11 (Experimental)
  Interventions: Drug: BMS-985521; Other: Placebo
- Part C (Experimental)
  Interventions: Drug: BMS-985521

INTERVENTIONS:
Drug: BMS-985521 — Specified dose on specified days.
Other: Placebo — Specified dose on specified days
  Arms: Part A Cohort 1; Part A Cohort 2; Part A Cohort 3; Part A Cohort 4; Part A Cohort 5; Part A Cohort 6; Part B Cohort 10; Part B Cohort 11; Part B Cohort 7; Part B Cohort 8; Part B Cohort 9

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and drug levels of BMS-986521 following single and multiple ascending doses of BMS-986521 in healthy adult participants, and to evaluate potential food effects on BMS-986521 exposure.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy males and females (assigned at birth) who are not of childbearing potential, with no clinically significant abnormalities in medical history, physical exam, ECG, or lab tests.
* Participants must have a body mass index (BMI) between 18 and 32 kg/m² (inclusive) and body weight of at least 50 kg.
* For Part B/Cohort 11 only: participants with stable cardiovascular conditions may be included if deemed suitable by the investigator.

Exclusion Criteria:

* Participants must not have any significant medical condition or history (renal, hepatic, hematologic, GI, endocrine, pulmonary, neurologic, or immunologic) that may affect drug absorption, distribution, metabolism, or excretion (ADME), or pose a risk to the participant.
* Participants must not have a history of rhabdomyolysis, cancer (except certain cured skin or cervical cancers), hematologic malignancy, or myelodysplastic syndrome.
* Participants must not have recent or current significant GI disease, major surgery, or medical interventions affecting ADME (except appendectomy or cholecystectomy).
* Participants must not have had a blood transfusion within 4 weeks or have an inability to tolerate oral medication or venous access.
* Other protocol defined inclusion/exclusion criteria apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2026-11-17 (Estimated); Study Completion 2026-11-17 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (AEs) | Up to approximately Day 40
Number of participants with treatment-emergent serious adverse events (SAEs) | Up to approximately Day 40
Number of participants with Treatment-emergent suicidal ideation and behavior as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to approximately Day 14

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) of BMS-986521 in Plasma | Up to approximately Day 14
Time to Cmax (Tmax) of BMS-986521 in Plasma | Up to approximately Day 14
Area Under the Concentration-Time Curve from Time Zero to the Last Measured Time Point (AUC(0-T)) of BMS-986521 in Plasma | Up to approximately Day 14
Area Under the Concentration-Time Curve from Time Zero to 24 Hours (AUC(0-24)) of BMS-986521 in Plasma | Up to approximately Day 14
Area Under the Concentration-Time Curve from Time Zero Extrapolated to Infinity (AUC(INF)) of BMS-986521 in Plasma | Up to approximately Day 14
Concentration Over a Dosing Interval (tau) (AUC(TAU)) of BMS-986521 in Plasma | Up to approximately Day 14
Elimination Half-Life (T-HALF) of BMS-986521 in Plasma | Up to approximately Day 14
Apparent Clearance of BMS-986521 from Plasma after Dosing (CLT/F) | Up to approximately Day 14
Apparent Volume of Distribution in Plasma after Dosing (Vz/F) of BMS-986521 | Up to approximately Day 14
Accumulation Index Based on Maximum Concentration (Cmax) in Plasma after Multiple Dosing (AI_Cmax) of BMS-986521 | Up to approximately Day 14
Accumulation Index Based on Area Under the Curve (AUC) in Plasma After Multiple Dosing (AI_AUC) of BMS-986521 | Up to approximately Day 14
Geometric Mean Cmax BMS-986521 under fed and fasted conditions | Up to approximately Day 11
  Cohort 3
Geometric Mean AUC(0-T) BMS-986521 under fed and fasted conditions | Up to approximately Day 11
  Cohort 3
Geometric Mean AUC(INF) BMS-986521 under fed and fasted conditions | Up to approximately Day 11
  Cohort 3
Geometric mean ratios of Cmax for BMS-986521 oral tablet vs solution | Up to approximately Day 11
  Part C
Geometric mean ratios of AUC(0-T) for BMS-986521 oral tablet vs solution | Up to approximately Day 11
  Part C
Geometric mean ratios of AUC(INF) for BMS-986521 oral tablet vs solution | Up to approximately Day 11
  Part C

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- CenExel ACT (Formerly Anaheim Clinical Trials; LLC), Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07283263.html